CLINICAL TRIAL: NCT03392558
Title: The Suitability of Two Skin Care Regimens in Moderate to Severe Facial Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burt's Bees Inc. (Industry)
Collaborators: Dermatology Consulting Services, High Point NC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DCS-25-17
Record Dates: First submitted 2017-12-27; First posted 2018-01-08 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-Based Sensitive Skin Regimen (Experimental): Burt's Bees Skin Care Regimen (Nature Based Sensitive Skin Regimen, NBSSR):
  1. Burt's Bees Sensitive Facial Cleanser (to be used day and night)
  2. Burt's Bees Sensitive Daily Moisturizing Cream (to be used in the day)
  3. Burt's Bees Sensitive Night Cream (to be used at night)
  Interventions: Other: Burt's Bees Skin Care Regimen
- Control Regimen (Active Comparator): Control Skin Care Regimen (Control Regimen, CR):
  1. Cetaphil Gentle Skin Cleanser (to be used day and night)
  2. Cetaphil Moisturizing Lotion (to be used day and night)
  Interventions: Other: Control Regimen

INTERVENTIONS:
Other: Burt's Bees Skin Care Regimen — Burt's Bees Facial Cleanser (twice daily), Burt's Bees Sensitive Daily Moisturizing Cream (morning), Burt's Bees Sensitive Night Cream (at bedtime)
  Arms: Nature-Based Sensitive Skin Regimen
Other: Control Regimen — Cetaphil Gentle Skin Cleanser (twice daily), Cetaphil Moisturizing Lotion (twice daily)
  Arms: Control Regimen

SUMMARY:
This study evaluates a nature-based sensitive skin regimen (NBSSR), as a suitable adjunct topical application to prescription medication when administered daily over the course of four weeks, in moderate to severe rosacea in comparison to the control regimen (CR).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be female 25-60 years of age with moderate facial rosacea at screening and 6 or 7 papules and/or pustules; as well as, no other known medical conditions that, in the investigator's opinion, may interfere with study participation.
* Women of childbearing potential must be willing to use a form of birth control during the study. For the purpose of this study, the following are considered acceptable methods of birth control: oral contraceptives, Norplant(R), Depo-Provera(R) double barrier methods (e.g., condom and spermacide) and abstinence.
* Subjects must provide written informed consent.
* Willingness to comply with the study design and procedures.
* Subjects who agree to sign a photography release form.

Exclusion Criteria:

* Any dermatological disorder, except rosacea requiring the use of prescription medication, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin characteristics,
* Subjects who are using any anti-aging skin care products within 4 weeks of study enrollment.
* Subjects who are not willing to use only the assigned study products and nothing else, except for self-selected colored cosmetics that must remain unchanged during the study, to their face.
* Subjects who have demonstrated a previous hypersensitivity reaction to any of the ingredients of the study products.
* Subjects, who are pregnant, breast feeding, or planning a pregnancy.
* Subjects with clinically significant unstable medical disorders.
* Subjects who are unwilling or unable to comply with the requirements of the protocol.
* Subjects who have history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study.
* Subjects who have participated in any clinical study in the past 30 days or are currently participating in any other clinical study.
* Subjects with any planned surgeries and/or invasive medical procedures during the course of the study.
* Subjects who started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.
* Subjects who currently or frequently use high doses of anti-inflammatory drugs for a defined medication condition. Aspirin use should not exceed 2 tablets (650 mg) per day.
* Subjects currently receiving any anticancer, immunosuppressive treatments/ medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.), or radiation as determined by the initial paperwork.
* Subjects with a history of immunosuppression/immune deficiency disorders (including (HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.) and/or radiation as determined by study documentation.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment of Rosacea Scale Score | 4 weeks
  The primary efficacy endpoint is no increase in the cumulative Investigator Global Assessment of Rosacea Scale score, measured at Week 4 from baseline

SECONDARY OUTCOMES:
Overall Skin Quality | 4 weeks
  The secondary efficacy endpoint is at least no increase in the Overall Skin Quality domain of the Subject-Rated Efficacy Scale score, measured at Week 4 from baseline

OTHER OUTCOMES:
Transepidermal Water Loss | 4 weeks
  No increase in transepidermal water loss values measured at Week 4 from baseline
Corneometry | 4 weeks
  No decrease in corneometry values at Week 4 from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zoe D Draelos, MD, Principal Investigator — Dermatology Consulting Services, High Point NC
Locations (1):
- Dermatology Consulting Services, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Draelos ZD, Gunt H, Levy SB. Natural Skin Care Products as Adjunctive to Prescription Therapy in Moderate to Severe Rosacea. J Drugs Dermatol. 2019 Feb 1;18(2):141-146. PMID 30794364